CLINICAL TRIAL: NCT07183111
Title: Comparison of Traditional Instructions Vs AI Based Instructions With Customized Chat GPT as Remote Support System on Education of Orthodontic Patients:A Randomised Control Trial
Brief Title: Comparison of Traditional Instructions Vs AI Based Instructions With Customized Chat GPT as Remote Support System on Education of Orthodontic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Syeda Ayesha Fatima, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SOD/ERB/2025/90
Record Dates: First submitted 2025-09-06; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Focus of the Study is Plaque and Gingival Index Score Before and After Instructions; Satisfaction Assessment of Orthodontic Patients With Both Instruction Modalities; Knowledge Assessment; Recall Ability of Orthodontic Instructions With Both Modalities
Keywords: AI in orthodontics; Chatbots and health education
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group:chat bot group (Experimental): Intervention group : receives instructions from advance voice feature of chat gpt chair side and customized chat gpt as home care remote support in form of chat bot
  Interventions: Other: Instructions given via artificial intelligence chatbot in form of voice instructions at chair side with Customized chatbot for remote home support
- Control group: traditional instructions chairside verbally with pamphlet support (Active Comparator): Control group : receives instructions verbally on chair side with pamphlet as home care remote support
  Interventions: Other: Control group instructions given by chair side orthodontist verbally and written pamphlet as home care support

INTERVENTIONS:
Other: Instructions given via artificial intelligence chatbot in form of voice instructions at chair side with Customized chatbot for remote home support — Instructions given via artificial intelligence chatbot in form of voice instructions at chair side with Customized chatbot for remote home support
  Arms: intervention group:chat bot group
Other: Control group instructions given by chair side orthodontist verbally and written pamphlet as home care support — Control group instructions given by chair side orthodontist verbally and written pamphlet as home care support
  Arms: Control group: traditional instructions chairside verbally with pamphlet support

SUMMARY:
This study will assess the impact of voice instructions delivered by advance voice feature of Chat gpt followed by remote support with chatbot in form of customized chat gpt named Brace AI which is customized by principal investigator.AI generate post operative instructions will be compared with post bracketing instructions given verbally in traditional chair side manner and home support with pamphlet in terms of oral hygiene outcome ,satisfaction with both modalities of instruction , recall ability and knowledge of the orthodontic patients

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-30 years undergoing bracket placement
* No prior experience of orthodontic treatment
* In good state of physical and mental health
* Understand the medium of instructions properly which will be Urdu language in this study
* Internally motivated patients with fairly good oral hygiene at the start of treatment
* Access to smart phone or internet at home

Exclusion Criteria:

* Systemic conditions affecting oral hygiene
* Cognitive impairments that may hinder comprehension
* Patients with language barriers that might affect their understanding of

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Plaque index | T0 at baseline T1 1 month T2 2 months T 3 3 months
  Score from O-3 0=no plaque 3=abundant plaque
Modified gingival index | T0 at baseline T1 1 month T2 2 months T 3 3 months
  Score from 0-4 0= normal gingival tissue 4=erythema edema gingival hypertrophy and spontaneous bleeding

SECONDARY OUTCOMES:
Knowledge assessment | T0 at baseline T1 at 1 month T2 at 2 months T3 AT 3 months
  Scale from 0-4 0=very little 4=excellent
Patient satisfaction with instruction modality | T0 at baseline T1 at 1 month T2 at 2 months T3 AT 3 months
  Measured with satisfaction scale 0-4 0=very unsatisfactory 4=very satisfactory
Recall ability | T0 at baseline T1 at 1 month T2 at 2 months T3 AT 3 months
  Measured via quiz

CONTACTS AND LOCATIONS:
Locations (1):
- School of dentistry Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sevgi M, Antaki F, Keane PA. Medical education with large language models in ophthalmology: custom instructions and enhanced retrieval capabilities. Br J Ophthalmol. 2024 Sep 20;108(10):1354-1361. doi: 10.1136/bjo-2023-325046. PMID 38719344
- [Background] Santonocito S, Cicciu M, Ronsivalle V. Evaluation of the impact of AI-based chatbot on orthodontic patient education: a preliminary randomised controlled trial. Clin Oral Investig. 2025 Apr 30;29(5):278. doi: 10.1007/s00784-025-06356-8. PMID 40304793

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-07-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT07183111/Prot_SAP_ICF_000.pdf